CLINICAL TRIAL: NCT02855463
Title: Study of Giant Viruses of Amoebas Infections in Children Suffering From Gastroenteritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_3755 - 1930
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Gastroenteritis
Keywords: Giant virus; Amoeba
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The discovery in 2003 by isolation of amoebas Mimivirus, the world's largest virus at the Research Unit on Tropical and Emerging Diseases in Marseille revealed fascinating information about the definition and evolution of viruses. Its genome encodes about 1,000 proteins. Three other viruses were then isolated from amoebas in this unit:Two other giant viruses, Mamavirus Marseillevirus then, and the first virus a virus, named virophage, which led to highlight the role of amoeba (Acanthamoeba spp. ) such as spawning giant viruses and compounds of bacterial origin or cellular proteins This project focuses on the detection and analysis of new viral agents (viruses and virophages giant amoeba environmental) and their involvement in human pathology.

The objectives of this study are observational: detect and document the presence of giant viruses and virophages of amoebae in the faeces of children presenting to the pediatric emergency reception service of the North Hospital in AP -HM with or without clinical evidence of gastroenteritis.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted in the Pediatric Emergency Service of Northern Hospital, Marseille, France
* Patient aged ≤ 15.3 years, male or female;
* Patient for whom a microbiological exam should be performed during the clinical management, with or without a clinical diagnosis of gastroenteritis (ie including diarrhea which will be defined by the issuance of at least three molded or watery stools per day for more than 24 hours) at the time of the collection of stool;
* Patient for whom informed consent was read, understood, signed by a parent or legal representative.

Exclusion criteria

* Patient aged > 15.3 years;
* Patient for whom informed consent is not signed by a parent or legal representative.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children admitted for gastroenteritis who need a microbiological exam to confirm diagnosis
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-07; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of children carriers in their digestive tract of giant viruses (and their virophages) associated with amoebae | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided